CLINICAL TRIAL: NCT04530747
Title: Metabolic Effects of Metformin Therapy in Obstructive Sleep Apnea
Acronym: MET-OSA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recall of positive airway pressure (PAP) device.
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Prachi Singh, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PBRC 2020-033; P30DK072476 (NIH)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Metformin
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin + PAP (Experimental): Subjects randomized to this arm will be orally given 2000 mg metformin daily. Metformin dosage will be slowly increased to improve tolerance.
  Subjects will also be provided PAP (positive airway pressure) device for standard management of obstructive sleep apnea.
  Interventions: Drug: Metformin + PAP
- Placebo oral capsule + PAP (Placebo Comparator): Subjects randomized to this arm will receive placebo matching study drug. Subjects will also be provided PAP (positive airway pressure) device for standard management of obstructive sleep apnea.
  Interventions: Drug: Placebo oral capsule + PAP

INTERVENTIONS:
Drug: Metformin + PAP — Subjects randomized to this arm will receive 500 mg capsules containing metformin extended release (XR). Metformin XR dosing will be 500 mg (1 x 500 mg) every evening (qPM) during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided PAP (positive airway pressure) device for standard management of obstructive sleep apnea.
  Arms: Metformin + PAP
Drug: Placebo oral capsule + PAP — Subjects randomized to this arm will receive 500 mg capsules containing placebo. Placebo dosing will be 500 mg (1 x 500 mg) qPM during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided PAP (positive airway pressure) device for standard management of obstructive sleep apnea.
  Arms: Placebo oral capsule + PAP

SUMMARY:
The purpose of the study is to see if metformin improves metabolism in patients with obstructive sleep apnea (OSA) using positive airway pressure (PAP) therapy. Metformin is approved by the Food and Drug Administration (FDA) for the treatment and prevention of diabetes. It is not approved for use in patients with OSA.

DETAILED DESCRIPTION:
Positive airway pressure (PAP) is standard therapy for obstructive sleep apnea (OSA) but has shown mixed results for improvement of insulin sensitivity and does not reduce cardiovascular (CV) events and mortality, even in patients with established CV disease. Hence, eliminating intermittent hypoxia alone with standard PAP therapy may not be sufficient to restore metabolism. Additional adjunct strategies (such as metformin) known to improve metabolism may be required to reduce metabolic burden and CV risk in OSA patients. The aim of this study is to examine the longitudinal changes in metabolism of OSA patients receiving both PAP and metformin treatment.

The MET-OSA study will last about 4 months. After screening the participants to determine eligibility, baseline study measures will be obtained and the participants will be provided with standard PAP for OSA treatment. Participants will also be randomized to receive either placebo or metformin treatment for 3 months. Compliance to study drug will be determined during monthly follow-up visits. Final study visit will include assessment of all baseline study measures.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 30-50 kg/m^2 (inclusive).
* Apnea-Hypopnea Index ≥ 15 events/h.
* Must be able to provide written informed consent.
* Willing to participate and adhere to study procedures (video recorded in-lab sleep studies, positive airway pressure (PAP) treatment, take study drug, have adipose tissue and skeletal muscle biopsies).
* Women of child-bearing potential must agree to use appropriate contraception to avoid pregnancy throughout the study.
* Willing to have blood, as well as adipose and muscle tissue stored for future use.

Exclusion Criteria:

* HbA1c > 6.4%.
* Severe or uncontrolled hypertension defined as systolic blood pressure (BP) ≥180 mmHg and/or diastolic BP ≥110 mmHg on the average of three seated measurements after being at rest for at least 5 minutes.
* Significant cardiovascular, hepatic, renal, neurologic, or psychiatric disease as determined by the study physician.
* Pregnancy, breast feeding or planning pregnancy in the coming 4 months.
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) <60ml/min/1.73m2 (estimated with Chronic Kidney Disease Epidemiology Collaboration equation 1 method).
* Known hypersensitivity to metformin.
* Currently taking a glucose lowering or weight loss medications.
* Current PAP use or use of PAP in the past 6 months.
* Currently taking antihypertensive and lipid-lowering medications known to affect adipose tissue and skeletal muscle metabolism. For example, statins and drugs targeting renin-angiotensin system will not be allowed. However, use of diuretics, beta-blockers, alpha-blockers and calcium channel blockers may be allowed provided the participant is on a stable dose for at least 3 months prior to the study visit.
* Oxygen desaturation index <15 events/h of sleep.
* Any medication or condition that, in the opinion of the medical investigator, could interfere with the study outcomes or put the subject at risk by participating in the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prachi Singh, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Recruiting core Pennington, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin + PAP: Subjects randomized to this arm will be orally given 2000 mg metformin daily. Metformin dosage will be slowly increased to improve tolerance.
  Metformin: Subjects randomized to this arm will receive 500 mg capsules containing metformin extended release (XR). Metformin XR dosing will be 500 mg (1 x 500 mg) every evening (qPM) during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided positive airway pressure (PAP) device for standard management of obstructive sleep apnea.
- Placebo Oral Capsule + PAP: Subjects randomized to this arm will receive placebo matching study drug.
  Placebo oral capsule: Subjects randomized to this arm will receive 500 mg capsules containing placebo. Placebo dosing will be 500 mg (1 x 500 mg) every evening (qPM) during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided positive airway pressure (PAP) device for standard management of obstructive sleep apnea.
Period: Overall Study
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metformin + PAP: Subjects randomized to this arm will be orally given 2000 mg metformin daily. Metformin dosage will be slowly increased to improve tolerance.
  Metformin: Subjects randomized to this arm will receive 500 mg capsules containing metformin XR. Metformin XR dosing will be 500 mg (1 x 500 mg) qPM during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided PAP (positive airway pressure) device for standard management of obstructive sleep apnea.
- Placebo Oral Capsule + PAP: Subjects randomized to this arm will receive placebo matching study drug.
  Placebo oral capsule: Subjects randomized to this arm will receive 500 mg capsules containing placebo. Placebo dosing will be 500 mg (1 x 500 mg) qPM during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided PAP (positive airway pressure) device for standard management of obstructive sleep apnea.
- Total: Total of all reporting groups
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.25 (8.31) | 51.5 (5.04) | 50.88 (6.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] | 36.63 (2.34) | 36.31 (3.48) | 36.47 (2.87)
Apnea Hypopnea Index [Mean (Standard Deviation); unit: event/h of sleep] — Apnea Hypopnea Index is the number of apneas (temporary cessation of breath) or hypopneas (shallow breathing) experienced per hour of sleep.
  event/h of sleep | 54.4 (22.5) | 52.1 (21) | 53.3 (21.1)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Matsuda Index
Description: Comparison of change in Matsuda Index as determined by 2-h oral glucose tolerance test (OGTT). During OGTT, response to oral 75g glucose intake is determined by measuring insulin and glucose in timed samples obtained at -5, 10, 20, 30, 60, 90 and 120 min. Matsuda index is a commonly used composite index to estimate whole-body insulin sensitivity. Matsuda index is calculated as (10,000/ square root of [fasting glucose X fasting insulin] X [mean OGTT glucose X mean OGTT insulin]). Increase in scores reflect improvement in whole body insulin sensitivity.
Time Frame: approximately 4 months, includes measures obtained at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP
Number analyzed (Participants) | 7 | 8
Index | 0.395 (1.695) | -0.649 (1.974)

2. Secondary Outcome: Changes in Insulin Area Under the Curve (AUC) During 2-h Oral Glucose Tolerance Test (OGTT)
Description: Comparison of change in insulin AUC (area under the curve) as derived from 2-h oral glucose tolerance test (OGTT). During OGTT, response to oral 75g glucose intake is determined by measuring insulin and glucose in timed samples obtained at -5, 10, 20, 30, 60, 90 and 120 min. 2-h insulin AUC is calculated using trapezoid method. Higher AUC indicates higher insulin secretion.
Time Frame: approximately 4 months, includes measures obtained at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: uU*120min/mL
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP
Number analyzed (Participants) | 7 | 8
uU*120min/mL | -855 (3334) | 4222 (4482)

3. Secondary Outcome: Changes in Glucose Area Under the Curve (AUC) During 2-h Oral Glucose Tolerance Test (OGTT)
Description: Comparison of change in glucose AUC (area under the curve) as derived from 2-h oral glucose tolerance test (OGTT). During OGTT, response to oral 75g glucose intake is determined by measuring insulin and glucose in timed samples obtained at -5, 10, 20, 30, 60, 90 and 120 min. 2-h glucose AUC is calculated using trapezoid method. Higher AUC indicates higher levels of circulating glucose.
Time Frame: approximately 4 months, includes measures obtained at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: mg*120min/dL
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP
Number analyzed (Participants) | 7 | 8
mg*120min/dL | -1759 (4260) | 698 (2754)

4. Secondary Outcome: Changes in Insulinogenic Index
Description: Comparison of insulinogenic index derived from the initial 30 min data from the 2-h oral glucose tolerance test (OGTT). Insulinogenic index measures the early insulin response during the oral glucose challenge. The index is calculated as ratio of change in insulin to glucose from 0 to 30 min values derived from OGTT. Decrease in scores reflect improvement in insulin sensitivity.
Time Frame: approximately 4 months, includes measures obtained at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP
Number analyzed (Participants) | 7 | 8
Index | 0.201 (0.497) | 0.206 (0.529)

5. Secondary Outcome: Changes in Disposition Index
Description: Comparison of change in disposition index as derived from 2-h oral glucose tolerance test. Disposition index measures beta-cell function and is calculated as product of Matsuda index and Insulinogenic index values. Increase in scores reflect improvement in glucose metabolism.
Time Frame: approximately 4 months, includes measures obtained at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Metformin + PAP: Subjects randomized to this arm will be orally given 2000 mg metformin daily. Metformin dosage will be slowly increased to improve tolerance.
  Metformin: Subjects randomized to this arm will receive 500 mg capsules containing metformin XR. Metformin XR dosing will be 500 mg (1 x 500 mg) qPM during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided positive airway pressure (PAP) device for standard management of obstructive sleep apnea.
- Placebo Oral Capsule + PAP: Subjects randomized to this arm will receive placebo matching study drug.
  Placebo oral capsule: Subjects randomized to this arm will receive 500 mg capsules containing placebo. Placebo dosing will be 500 mg (1 x 500 mg) qPM during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
  Subjects will also be provided positive airway pressure (PAP) device for standard management of obstructive sleep apnea.
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP
Number analyzed (Participants) | 7 | 8
Index | 0.617 (1.357) | -0.012 (1.726)

6. Secondary Outcome: Changes in Homeostasis Model Assessment for Insulin Resistance (HOMA-IR)
Description: Comparison of change in HOMA-IR value derived from fasting insulin and glucose. HOMA-IR is a simple index for insulin resistance based on fasting measures of glucose and insulin which is a commonly used end-point for assessment of insulin resistance in clinical trials. HOMA-IR is calculated as [(fasting insulin X fasting glucose)/ 22.5]. Higher values indicate higher insulin resistance. An increase will suggest a detrimental effect on glucose metabolism. Individuals with HOMA-IR < 5.7% are considered healthy, between 5.7 and 6.4% are considered prediabetic, and more than 6.4% are considered diabetic.
Time Frame: approximately 4 months, includes measures obtained at baseline and 3 month follow-up.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Metformin + PAP | Placebo Oral Capsule + PAP
Number analyzed (Participants) | 7 | 8
Index | 0.651 (2.274) | 1.981 (3.406)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Metformin: Subjects randomized to this arm will be orally given 2000 mg metformin daily. Metformin dosage will be slowly increased to improve tolerance.
  Metformin: Subjects randomized to this arm will receive 500 mg capsules containing metformin XR. Metformin XR dosing will be 500 mg (1 x 500 mg) qPM during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
- Placebo Oral Capsule: Subjects randomized to this arm will receive placebo matching study drug.
  Placebo oral capsule: Subjects randomized to this arm will receive 500 mg capsules containing placebo. Placebo dosing will be 500 mg (1 x 500 mg) qPM during Week 1, 1000 mg (2 x 500 mg) qPM during Week 2, 1500 mg (3 x 500 mg) qPM during Week 3, and 2000 mg (4 x 500 mg) qPM from Week 4 onwards.
Arm/Group | Metformin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Early termination due to PAP recall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT04530747/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT04530747/ICF_001.pdf